CLINICAL TRIAL: NCT04772105
Title: Phase Ib/IIa Clinical Study of the Safety and Efficacy of BAT5906 Injection in Patients With Diabetic Macular Edema With Multiple Changes of Intravitreal Two Doses
Brief Title: Clinical Study of the Safety and Efficacy of BAT5906 Injection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAT5906-003-CR
Record Dates: First submitted 2020-06-22; First posted 2021-02-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Intervention Model Description: one investigational medicine with two different dose groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.5mg of BAT5906 (Experimental): Specification: 10mg/0.2ml/piece; route of administration: intravitreal injection; dose: 2.5mg/eye/time, 50μl; medication duration: once every 4 weeks, 6 consecutive times, then every 4 weeks Followed up once (the investigator judged to administer the drug as needed) and observed until the 48th week.
  Interventions: Drug: 2.5mg of BAT5906
- 4mg of BAT5906 (Experimental): Specification: 16mg/0.2ml/piece; route of administration: intravitreal injection; dose: 4mg/eye/time, 50μl; medication duration: once every 4 weeks, 3 consecutive times, then every 4 weeks Followed up once (the investigator judged to administer the drug as needed) and observed until the 48th week.
  Interventions: Drug: 4.0mg of BAT5906

INTERVENTIONS:
Drug: 2.5mg of BAT5906 — Specification: 2.5mg of BAT5906
  Arms: 2.5mg of BAT5906
Drug: 4.0mg of BAT5906 — Specification: 4.0mg of BAT5906
  Arms: 4mg of BAT5906

SUMMARY:
This study is a multi-center, open, multiple-dose phase Ib/IIa clinical study evaluating the efficacy and safety of BAT5906 injection in patients with diabetic macular edema. BAT5906's phase I study on w-AMD shows that it is safe from 0.3-4.0 mg, and the higher dose (2.5 mg and 4 mg) may maintain the effect for longer; the same target drugs (such as brolucizumab and Abecip ) It has also been found in clinical studies that high doses can extend the dosing interval and reduce the dosing frequency. Therefore, in this study, two safe and effective doses were selected, and the optimal clinical effective dose and frequency of BAT5906 in DME were initially explored.

ELIGIBILITY:
Inclusion Criteria:

* Only the following criteria are met:

  1. Sign the informed consent voluntarily, willing and capable to follow the procedures of outpatient visits and research at the time specified in the trial
  2. Diagnosed with type 1 or type 2 diabetes, aged 18 to 80 years old;
  3. The drug treatment to control diabetes must be stable within 3 months before randomization and is expected to remain stable during the study period;
  4. Macular edema secondary to diabetes, and found to be involved in the macular center (fovea) of the research eye by OCT examination, confirmed by the reading center during screening;
  5. The CRT of the research eye evaluated by OCT examination is ≥300 μM, confirmed by the reading center during screening;
  6. The BCVA of the research eye is 73-24 letters (using the ETDRS table, including the boundary value, which is equivalent to the Snellen visual acuity score of the research eye equal to 20/40 -20/400);
  7. Contralateral eye BCVA ≥ 34 letters (using ETDRS table, equivalent to snellen vision ≥ 20/200). Note: If both eyes meet the inclusion criteria, the eye with poor baseline vision is selected as the research eye;
  8. At the time of screening and baseline, the investigator judged that the contralateral eye was expected to not require any anti-VEGF treatment within 3 months (PK group only).

Exclusion Criteria:

* If a patient meets any of the following conditions, they cannot enter the study:

Eye exclusion criteria:

1. There is structural damage to the center of the macula in the eye, and the best corrected vision may not be improved after the macular edema resolves, including atrophy of retinal pigment epithelial cells, subretinal fibrosis or scarring, and obvious macular ischemia (FFA suggests arching Obvious damage), macular anterior membrane involving fovea or organic hard exudate (as confirmed by the reading center before randomization);
2. The research eye has iris lesions and neovascular glaucoma;
3. Those who have no eye lens (except intraocular lens);
4. The study eye has active hyperplastic diabetic retinopathy (PDR);
5. The research eye has anyone other than diabetic macular edema that may confuse macular assessment or vision testing (retinal vascular occlusion, retinal detachment, vitreous macular traction, macular hole, preretinal fibrosis involving the macula, choroidal neovascularization, age Related macular degeneration, etc.);
6. The research eye is accompanied by poorly controlled glaucoma, which is defined as the intraocular pressure still ≥21mmHg after treatment with anti-glaucoma drugs, or according to the judgment of the investigator;
7. The research eye has undergone or may have undergone anti-glaucoma surgery during the study period (including trabeculectomy, sclerectomy and non-penetrating trabecular surgery, etc.);
8. The research eye has undergone vitreoretinal surgery or scleral buckling;
9. At the time of screening and baseline, the study eye had received laser photocoagulation (total retina or macular laser photocoagulation) within 90 days (including 90 days) or during the study period;
10. At the time of screening and baseline, the study eye had any intraocular or perocular surgery within 90 days (including 90 days) (except for yttrium-aluminum-garnet (YAG) lens capsule incision and eyelid surgery for more than 30 days) ;
11. A history of uveitis in any eye;
12. Any eye has active ocular inflammation or infection (bacterial, viral, parasitic or fungal infection);
13. At the time of screening and baseline, any eye had received intraocular anti-VEGF treatment within the first 90 days (including 90 days), such as ranibizumab, bevacizumab, abercept, compacept, etc.;
14. At the time of screening and baseline, any eye has received intraocular, periocular, and subconjunctival corticosteroid treatment within the first 90 days (including 90 days);

    Exclusion criteria for abnormal conditions in laboratory inspection:
15. Abnormal liver and kidney function (this test specifies that ALT and AST should not be higher than the upper limit of the normal value of the laboratory in the center by 2.5 times; Crea and BUN should not be higher than the upper limit of the normal value of the laboratory in the center by 2 times);
16. Abnormal blood coagulation function (prothrombin time ≥ upper limit of normal value 3 seconds, activated partial thromboplastin time ≥ upper limit of normal value 10 seconds);
17. Any one of the infected patients: active hepatitis B (if HBsAg(+) requires HBV DNA must be> 500 IU/mL or the hospital maximum limit), hepatitis C, AIDS or syphilis (positive RPR test);

    Other exclusion criteria:
18. Myocardial infarction or stroke occurred within 6 months before the first dose;
19. Poorly controlled diabetes [defined as glycated hemoglobin (HbA1c)>9%)];
20. Accompanied by uncontrollable hypertension (defined as blood pressure >150/100 mmHg after treatment with antihypertensive drugs);
21. Patients who took large doses of oral or injectable corticosteroids and other hormonal drugs (>10 mg prednisolone or the same dose/day) within 6 months before screening, but patients who used steroid drugs for inhalation, nasal cavity or local skin small doses except;
22. Those who have undergone surgery within 1 month and have not healed, or according to the investigator's judgment;
23. There is a history of contraindications to the study drug, metabolic dysfunction, physical examination results, or a disease or symptom that is reasonably suspected of being based on clinical laboratory results is a contraindication to the study drug, which may affect the judgment of the study results, or make the subject suffer Higher risk of complications;
24. Allergy or contraindications to known research drugs or their ingredients, fluorescein or povidone iodine;
25. Those who participated in clinical trials of any drugs (except vitamins and minerals) or devices 90 days before the first dose (including 90 days);
26. Women who are pregnant, pregnant or breastfeeding (pregnancy is defined as a positive blood/urine pregnancy test in this trial); male or female subjects of fertility do not agree to the entire study period and within 3 months after the end of the visit period Take appropriate contraceptive measures (such as IUD, birth control pills or condoms, etc.). For women who have not been menopausal or have been menopausal but have not met the menopause time continuously for more than 12 months, and have not undergone sterilization surgery (ovarian and/or hysterectomy), they are defined as having fertility. The definition of fertility may be adjusted according to local standards in each region.

    Note: High-efficiency contraception methods include total abstinence, IUD, double barrier method (eg condom + diaphragm with spermicides, implanted contraceptives, hormonal contraceptives [contraceptives, implanted contraceptives, transdermal Patches, hormone-vaginal devices or sustained-release injections], or the partner has undergone a vasectomy and is confirmed to have no sperm);
27. The researchers believe that there are other conditions that need to be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Vital signs（ body temperature） | After patient resting for more than 3 minutes
  the patient's body temperature (axillary temperature) Any clinically significant abnormality should be reported as an adverse event and recorded in the original
Vital signs（heart rate/pulse） | After patient resting for more than 3 minutes
  heart rate/pulse Any clinically significant abnormality should be reported as an adverse event and recorded in the original
Vital signs（respiratory rate） | After patient resting for more than 3 minutes
  respiratory rate Any clinically significant abnormality should be reported as an adverse event and recorded in the original
Vital signs（blood pressure） | After patient resting for more than 3 minutes
  blood pressure Any clinically significant abnormality should be reported as an adverse event and recorded in the original
physical examination | The investigator or other authorized and qualified investigator shall perform the prescribed physical examination according to the evaluation schedule. During the visit, the investigator performed a physical examination as indicated by symptoms
  Physical examination should include at least general conditions, head and face, skin, lymph nodes, ears, nose, throat, respiratory system, cardiovascular system, abdomen (including liver and spleen), genitourinary system, musculoskeletal system, nervous system, and mental condition
laboratory examination（blood routine） | Screening period，Week 12, Week 24, Week 48 of the last visit
  In the test process will be carried out in accordance with the testing program flow chart of blood routine, the laboratory testing results of the subjects to evaluate the change of relative to the baseline, the each evaluate clinical significance of abnormal experimental value, the researchers don't think with basic diseases related to abnormal subjects as AE record
laboratory examination（outine urine） | Screening period，Week 12, Week 24, Week 48 of the last visit
  In the test process will be carried out in accordance with the testing program flow chart of routine urine , the laboratory testing results of the subjects to evaluate the change of relative to the baseline, the each evaluate clinical significance of abnormal experimental value, the researchers don't think with basic diseases related to abnormal subjects as AE record
laboratory examination（blood biochemical examination） | Screening period，Week 12, Week 24, Week 48 of the last visit
  In the test process will be carried out in accordance with the testing program flow chart of blood biochemical examination, the laboratory testing results of the subjects to evaluate the change of relative to the baseline, the each evaluate clinical significance of abnormal experimental value, the researchers don't think with basic diseases related to abnormal subjects as AE record
laboratory examination（blood coagulation function） | Screening period，Week 12, Week 24, Week 48 of the last visit
  In the test process will be carried out in accordance with the testing program flow chart of blood coagulation function, the laboratory testing results of the subjects to evaluate the change of relative to the baseline, the each evaluate clinical significance of abnormal experimental value, the researchers don't think with basic diseases related to abnormal subjects as AE record
electrocardiogram（12- Lead ECG） | Screening period of the first visit: Week 12 of the fifth visit, Week 24 of the eighth visit, and Week 48 of the last visit
  During the trial, the examination of the electrocardiogram (ecg) method must be consistent, and to evaluate the clinical significance of the results, will any researchers to make judgment for clinical significance of abnormal as adverse events were reported, and recorded in the original records and case report form, the subjects in the process of the entire study if there is clinical indications by researchers to determine whether the need for ecg examination.
anti-drug antibody (ADA) | 24 hours before 1, 2, 3, 4 dosing, 5 dosing to last visit, each dosing before and 24 hours before the last visit as needed
  Plasma samples for anti-drug antibody (ADA) detection were collected to detect the positive incidence of ADA associated with plasma levels of BAT5906
ocular and non-ocular adverse events (AE) and serious adverse events (SAE) | Adverse events were collected from the time the patient signed the informed consent to the time 28 days after the last dication
  Any adverse medical event that occurs after a subject participates in a clinical trial and receives the investigational drug, but is not necessarily cause-and-effect with the treatment.
  An adverse event can be any adverse or unexpected sign (including abnormal laboratory tests), symptom, or disease, whether or not it is drug related.

SECONDARY OUTCOMES:
Effectiveness evaluation | Week 24
  Main efficacy indicators (study eye) At week 24, Change in BCVA from baseline
  At week 24, the mean change of BCVA from baseline.
  Secondary efficacy indicators (research eyes):
  At 12th and 48th week, the mean change of BCVA from baseline; At week 12, week 24 and week 48, the average change of CRT from baseline after OCT examination; At Week 12, 24 and 48, the proportion of subjects whose BCVA increased ≥10 letters from baseline, BCVA increased ≥15 letters from baseline, and BCVA decreased ≥15 letters from baseline; The average number of BAT5906 injections in 24 weeks and 48 weeks. The definition of CRT is: the average thickness of the central retina with the fixation point as the center and a diameter of 1 mm.
Effectiveness evaluation | Week 12 and 48
  Secondary efficacy indicators (study eye) At week 12 and 48, the mean change of BCVA from baseline.
Effectiveness evaluation | at weeks 12, 24, and 48
  Changes in CRT from baseline were examined by OCT CRT:The mean thickness of the central retina with a diameter of 1mm, centered on the fixed point of view
Effectiveness evaluation | at weeks 12, 24, and 48
  Percentage of subjects whose BCVA increased by ≥10 letters from baseline, increased by ≥15 letters from baseline, and decreased by ≥15 letters from baseline;
Effectiveness evaluation | 24 weeks and 48 weeks
  Average number of injections for BAT5906

OTHER OUTCOMES:
Pharmacokinetic (PK) evaluation | Once within 24 hours before administration.6 hours after administration, 24 hours after administration (once every 3 days) up to 672 hours after administration
  Each treatment group collected blood samples throughout the study to detect the blood sample concentration of BAT5906 injection.
Peripheral blood VEGF evaluation (VEGF) | Once within 24 hours before administration.24 hours after administration (once every 7 days) up to 672 hours after administration
  Each treatment group collected blood samples throughout the study to detect blood VEGF concentration. Please refer to the PK/VEGF/ADA blood collection schedule for the collection time of peripheral VEGF blood samples.
  Evaluation index: change level of peripheral blood VEGF before and after administration
Evaluation of immunogenicity | First administration: within 24 hours prior to administration.168 hours and 336 hours after administration, and the second until the last administration: within 24 hours before administration
  Detection of anti-BAT5906 antibody (ADA), please refer to PK/VEGF/ADA blood collection timetable for blood sample collection time. Detection of anti-drug antibody (ADA) in serum, if the ADA confirmed positive samples will continue to neutralize antibody (Nab) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College
Locations (19):
- China (19):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijiang, Beijing Municipality
  - Eye Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Henan Provincial Eye Hospital, Henan
  - Jieyang People's Hospital, Jieyang
  - The First Hospital of Jilin University, Jilin
  - The Affiliated Eye Hospital of Nanchang University, Nanchang
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Affiliated Hospital of Qingdao University, Qingdao
  - Joint Shantou International Eye Center of Shantou University and The Chinese University of Hong Kong, Shantou
  - West China Hospital of Sichuan University, Sichuan
  - Wenzhou Medical University Affiliated Optometry Hospital, Wenzhou
  - The Second Xiangya Hospital of Central South University, Xiangya
  - Xiangya Hospital Central South University, Xiangya
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou